CLINICAL TRIAL: NCT06523335
Title: Intermuscular Coordination as a Novel Clinical Target for Stroke Neurorehabilitation
Brief Title: Improving Independent Multi-joint Arm Control After Stroke
Acronym: NICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: UT Health Houston (Unknown); Korea Advanced Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Jinsook Roh, Assistant Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001333
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Muscle synergy; Intermuscular Coordination; Electromyogram-guided exercise; Motor neurorehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular coordination-guided rehabilitative training (Experimental): Post-stroke participants will perform a center-out task by generating isometric contractions of multiple muscles to move the cursor on a screen while electromyographic (EMG) responses are recorded. Activation of each muscle (or muscle group) will be mapped to 1 of 4 directions within the multi-dimensional cursor space. We will derive the cursor position in real time using EMGs recorded from multiple arm muscles.
  Interventions: Other: Neuromuscular coordination-guided rehabilitative training
- Force strengthening-guided rehabilitative training (Active Comparator): Post-stroke participants will perform a center-out task by generating isometric force to move the cursor on a screen. Participants will generate isometric force, which will move their cursor on the monitor. They will be trained to match one of the four force targets on display. We will derive the cursor position in real time using three forces (Fx, Fy, and Fz) measured at the load cell.
  Interventions: Other: Force strengthening-guided rehabilitative training

INTERVENTIONS:
Other: Neuromuscular coordination-guided rehabilitative training — During training exercise, post-stroke participants will be asked to match the targets on the screen. The experimental group will match them by activating a specific set of muscle. During assessment trials, a physical therapist or occupational therapist will rate the functional level of arm impairment using FMA and ARAT.
  Arms: Neuromuscular coordination-guided rehabilitative training
Other: Force strengthening-guided rehabilitative training — During training exercise, post-stroke participants will be asked to match the targets on the screen. The active comparator group will match them by generating isometric force in a desired target direction. During assessment trials, a physical therapist or occupational therapist will rate the functional level of arm impairment using FMA and ARAT.
  Arms: Force strengthening-guided rehabilitative training

SUMMARY:
The purposes of this study include:

1. - To identify whether features of aberrant intermuscular coordination patterns can be used to predict motor impairment after stroke.
2. - To test whether muscle synergies are malleable to a non-invasive EMG-guided exercise that induces changes in intermuscular coordination of upper extremity muscles after stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability in the United States. Of the more than 700,000 Americans who experience a stroke each year, two-thirds survive. 69% of patients who were admitted to a rehabilitation unit following stroke have mild to severe upper extremity dysfunction. Currently, there are more than seven million stroke survivors in the U.S., many of whom have long-term motor and sensory impairments, especially in the arm. The objective of this study involves both scientific and clinical aspects:

For the first purpose, intermuscular coordination patterns emerging under isometric reaching and dynamic conditions will be identified to predict impairment of both non-motion or motion-involved task performance and severity of motor impairment after stroke. This aim will enroll 15 age-matched (age of 40-75 yo) healthy adults and 25 adult (age of 40-75 yo) stroke survivors. Each stroke participant will have two visit sessions while age-matched will have a single measurement session.

For the second purpose, in total, 74 stroke survivors will perform an electromyographic signal-guided exercise through human-machine interaction to ameliorate motor impairment post-stroke by normalizing abnormal intermuscular coordination patterns in the arm after stroke, and improve motor impairment; also, assessment of the intermuscular coordination, UE Fugl-Meyer (FM), and Action Research Arm Test (ARAT) will be performed. Participants will have three visits per week for six weeks for training sessions. Finally, to test retention of the intervention effect, they will perform two assessment sessions one and three months after finishing the training.

ELIGIBILITY:
Inclusion criteria for aged matched healthy group

* Male or female whose age range between 40 and 75
* no known neurological injuries

Exclusion criteria for aged matched healthy group

* have an orthopedic disorder involving upper limbs;
* have a history of any neurologic disease;
* have any history of epilepsy of the potential participants and/or their family members;
* are unable to consent;
* are pregnant.

Inclusion criteria for stroke group

* male or female hemiparetic chronic stroke survivors;
* age ranging between 40-75 year;
* with single unilateral ischemic or hemorrhagic middle cerebral artery stroke;
* neurologically stable for >6 months;
* have an expectation that current medication will be maintained without changes for at least 3 months. Stable use of anti-spasticity medication (e.g., baclofen, diazepam, tizanidine) is accepted;
* without severe spasticity (Modified Ashworth (MA) <4);
* have not received botulinum toxin on the impaired arm within 3 months.

Exclusion criteria for stroke group

* have an orthopedic disorder involving upper limbs;
* cognitive impairment sufficient to interfere with informed consent or successful completion of the protocol (Montreal Cognitive Assessment (MoCA) score < 26);
* a history of another neurologic disease;
* anesthesia of joint position sense in upper limbs;
* are pregnant or have a chance that they might be (self-reported);

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) score | before any training, after the 6 weeks of training, respectively, and 1 and 3 months after the last training session, respectively
  To measure severity of motor impairment after stroke, FMA will be performed in the human upper extremity. FMA is commonly used to assess severity of motor impairment and motor recovery. The maximum FMA upper extremity motor score is 66 (i.e., 0: complete motor impairment; 66: normal motor performance). Each item is scored on a 3-point scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).
Change in Action Research Arm Test (ARAT) score | before any training, after the 6 weeks of training, respectively, and 1 and 3 months after the last training session, respectively
  To measure motor function after stroke, ARAT will be performed in the human upper extremity. 19 Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch, and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally).
Change in intermuscular coordination patterns | before any training, after the 6 weeks of training, respectively, and 1 and 3 months after the last training session, respectively
  EMGs will be recorded from 12 muscles. To assess whether muscle-synergy guided and/or force-guided exercise induce changes in the composition of intermuscular coordination patterns, non-negative matrix factorization will be applied to EMGs to identify and compare ICoPs.

SECONDARY OUTCOMES:
Brain imaging data recording | before any training, after the 6 weeks of training, respectively, and 1 and 3 months after the last training session, respectively
  A non-invasive electroencephalography (EEG) measurement setup will be employed to collect the EEG signal, specifically, thirty-two EEG electrodes will be placed on the scalp, and EEG signals will be measured during an isometric assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsook Roh, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thom T, Haase N, Rosamond W, Howard VJ, Rumsfeld J, Manolio T, Zheng ZJ, Flegal K, O'Donnell C, Kittner S, Lloyd-Jones D, Goff DC Jr, Hong Y, Adams R, Friday G, Furie K, Gorelick P, Kissela B, Marler J, Meigs J, Roger V, Sidney S, Sorlie P, Steinberger J, Wasserthiel-Smoller S, Wilson M, Wolf P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2006 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2006 Feb 14;113(6):e85-151. doi: 10.1161/CIRCULATIONAHA.105.171600. Epub 2006 Jan 11. No abstract available. PMID 16407573
- [Background] Parker VM, Wade DT, Langton Hewer R. Loss of arm function after stroke: measurement, frequency, and recovery. Int Rehabil Med. 1986;8(2):69-73. doi: 10.3109/03790798609166178. PMID 3804600
- [Background] Dewald JP, Pope PS, Given JD, Buchanan TS, Rymer WZ. Abnormal muscle coactivation patterns during isometric torque generation at the elbow and shoulder in hemiparetic subjects. Brain. 1995 Apr;118 ( Pt 2):495-510. doi: 10.1093/brain/118.2.495. PMID 7735890
- [Background] Roh J, Rymer WZ, Beer RF. Robustness of muscle synergies underlying three-dimensional force generation at the hand in healthy humans. J Neurophysiol. 2012 Apr;107(8):2123-42. doi: 10.1152/jn.00173.2011. Epub 2012 Jan 25. PMID 22279190
- [Background] Roh J, Rymer WZ, Perreault EJ, Yoo SB, Beer RF. Alterations in upper limb muscle synergy structure in chronic stroke survivors. J Neurophysiol. 2013 Feb;109(3):768-81. doi: 10.1152/jn.00670.2012. Epub 2012 Nov 14. PMID 23155178
- [Background] Carpinella I, Lencioni T, Bowman T, Bertoni R, Turolla A, Ferrarin M, Jonsdottir J. Effects of robot therapy on upper body kinematics and arm function in persons post stroke: a pilot randomized controlled trial. J Neuroeng Rehabil. 2020 Jan 30;17(1):10. doi: 10.1186/s12984-020-0646-1. PMID 32000790
- [Background] Wright ZA, Rymer WZ, Slutzky MW. Reducing Abnormal Muscle Coactivation After Stroke Using a Myoelectric-Computer Interface: A Pilot Study. Neurorehabil Neural Repair. 2014 Jun;28(5):443-51. doi: 10.1177/1545968313517751. Epub 2013 Dec 27. PMID 24376069
- See also: Laboratory Webpage — https://www.reignlaboratory.com/projects-3